CLINICAL TRIAL: NCT06634758
Title: The Effect Of Nursing Care Based On Watson's Human Care Model On Quality Of Life Of Patients iıth Multıple Sclerosis
Brief Title: The Effect of the Human Care Model on Patients With Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: a3xktrbv
Record Dates: First submitted 2024-09-17; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2023-10

CONDITIONS: Nursing Caries
Keywords: Nursing Care; Multiple Sclerosis; Quality of Life; Watson human care model
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Intervention Group Procedure 4 interviews were conducted with patients in this group and in each interview, patients were given MS Symptom Management and Relaxation Exercise training. Nursing care based on the Human Care Model was provided.
  Control Group Procedure No intervention other than routine treatment and care was applied to the patients in the control group. Data Collection Form, MS Quality of Life Scale were applied to the patients. Face-to-face interviews were conducted with these patients two and a half months after the first interview and the MS Quality of Life Scale was applied again. After the study ended, between June and November 2023, Watson Human Care Model Based Nursing Care was applied to the patients in this group (1 patient could not attend the planned interviews due to a change of province and 1 patient could not take leave from work).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- "intervention" (Experimental): When the studies in the literature are examined, it has been presented that nursing care based on Watson's Human Caring Model increases the quality of life in various diagnosed patient groups, reduces depression and pain, increases sleep quality and provides glycemic control . However, to our knowledge, no research has been conducted on individuals with MS based on Watson's Human Caring Model. Based on the idea that the model to be used will cause a positive change in the quality of life of MS patients, it is anticipated that this model-based research, which is preferred, can guide the treatment, support and counseling services that nurses provide to MS patients and strengthen nursing care.
  Interventions: Behavioral: Nursing interventions based on the Watson Human Caring Model

INTERVENTIONS:
Behavioral: Nursing interventions based on the Watson Human Caring Model — In the literature review, it was noticed that nursing care based on the Watson Human Caring Model was applied to various patient groups but not to patients with MS.

SUMMARY:
Purpose: This study was conducted to determine the effect of nursing care based on Watsons Human Caring Model on the quality of life of patients with MS.

Materials and Methods: This randomized controlled study was conducted in Gülhane Training and Research Hospital, Neurology Department Outpatient Clinic between January and November 2023.Patients were assigned to groups according to block randomization. The study was conducted with a total of 74 patients, 37 in the intervention and 37 in the control group. Four interviews were conducted with the patients, and a nursing care protocol based on the Watson Human Caring Model was applied. Patients in the control group underwent routine procedure. The "Multiple Sclerosis Symptom Management Booklet" and "Relaxation Exercises" educational materials used in the study were evaluated with the DISCERN measurement tool and the written materials evaluation form. Research data were obtained using the Data Collection Form, MS Quality of Life Scale, Watson Patient Satisfaction Form and Semi-Structured Interview Form.

Keywords: Watson Human Caring Model, MS, nursing care, quality of life.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is a chronic disease that usually affects young adults, progresses with attacks and remissions, causes widespread demyelinating lesions in the central nervous system, and can lead to functional limitations, disability, or a decrease in quality of life. It is reported that the number of individuals diagnosed with MS is approximately 58 thousand in our country and more than 2.9 million worldwide. This means that one person is diagnosed with MS every five minutes worldwide. According to the data of the Turkish Statistical Institute , MS ranks sixth among causes of death in 2022 with 3.5% and first among diseases that cause disability . According to TUİK data, 153 people died due to MS in 2021 and 138 people died in 2022 . As can be understood from the high rates of disability and death, MS is an important disease that critically affects people&amp;#39;s lives and quality of life. MS usually begins with attacks due to demyelination of axons in the brain, optic nerve and spinal cord; over time, it turns into a neurodegenerative disease associated with lack of neurotrophic support and neuron loss. Depending on the location and degree of degeneration of sensory and/or motor neurons during the course of the disease, various neurological disorders such as gait disturbance, loss of balance, muscle strength loss, fatigue, cognitive impairment and sensory loss occur alone or together. The physical, psychosocial and cognitive deficiencies caused by all these disorders and the chronic course of the disease limit the individuals; participation in activities and social life in their daily lives, causing the patients, physical performance, social roles and quality of life to be negatively affected. It is important to ensure the physical, social and psychological well-being of individuals diagnosed with MS, to increase their quality of life and to ensure their active and healthy participation in economic and social life. Considering the characteristics of MS disease, factors such as being chronic and irreversible, progressing with attacks, uncertainty in the treatment and disease process, and side effects of the drugs used negatively affect the physical and psychological health of individuals. In the health service to be provided to individuals diagnosed with MS, it is necessary to work on new methods and techniques in addition to medical approaches. It is important to provide holistic nursing care to MS patients, which includes not only symptom treatment but also the psychosocial status of the patient and addresses the patients problems from every aspect. Holistic nursing care, which addresses the patient problems from every aspect, forms the basis of the Human Care Model of nursing theorist Jean Watson. For Watson, nursing care is a professional, aesthetic, moral and scientific interpersonal process with the interaction of two individuals in terms of physical, spiritual, sociocultural and mental aspects. Watsons Human Care Model consists of the common sharing of core values in interaction and trust, disease prevention and health promotion, teaching-learning, holistic-alternative help practices, the individuals free will and autonomy-autonomy, the harmony of emotional and spiritual needs and scientific problem solving in decision making. The Human Caring Model values holistic practices by considering the concepts of soul-body-mental as a whole. When the studies in the literature are examined, it has been presented that nursing care based on Watsons Human Caring Model increases the quality of life in various diagnosed patient groups, reduces depression and pain, increases sleep quality and provides glycemic control. However, to our knowledge, no research has been conducted on individuals with MS based on Watsons Human Caring Model. Based on the idea that the model to be used will cause a positive change in the quality of life of MS patients, it is anticipated that this model-based research, which is preferred, can guide the treatment, support and counseling services that nurses provide to MS patients and strengthen nursing care.

Purpose of the Study This study is to determine the effect of nursing care based on Watsons Human Caring Model on the quality of life of patients with MS.

Hypotheses of the Study H0: Nursing care based on Watsons Human Caring Model has no effect on the quality of life of MS patients.

H1: Nursing care based on Watsons Human Caring Model has an effect on the quality of life of MS patients.

ELIGIBILITY:
Inclusion Criteria:

* Having a score between 3-7 on the Expanded Disability Status Scale (EDSS) (Puz et al., 2018) divided the patients into two groups as EDSS<3 and EDSS≥3 and reported that the frequency of comorbidity was high in patients with EDSS scores of 3 and above. For this reason, patients with EDSS scores below 3 were not included in the study. In addition, patients with EDSS scores above 7 are dependent on the caregiver/helper. Since the quality of life of dependent patients may be affected by the caregiver, patients with EDSS scores above 7 were not included in the study).

  * Being between the ages of 18 and 65
  * Being able to speak and understand Turkish, not having a speech-comprehension disorder

Exclusion Criteria:

* Having an attack during the research process

  * Becoming pregnant during the research process
  * Not being able to attend any or more of the four planned meetings in line with the care plan based on the Watson Human Care Model created for this research
  * Wanting to leave the research

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-10-28 (Estimated); Study Completion 2024-11-28 (Estimated)

PRIMARY OUTCOMES:
Multiple Sclerosis Quality of Life (MSQOL)-54 scale | 10 weeks
  The effect of nursing care on quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Fatma İlknur ÇINAR, Prof. Dr., Study Director — SBÜ Gülhane Hemşirelik Fakültesi
Locations (1):
- Atatürk Sanatoryum Eğitim ve Araştırma Hastanesi, Ankara, Keçiören, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I do not prefer this work to be shared.

DOCUMENTS (1):
  • Informed Consent Form (2023-05-15): https://cdn.clinicaltrials.gov/large-docs/58/NCT06634758/ICF_000.pdf